CLINICAL TRIAL: NCT06247670
Title: A Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study of CMP-CPS-001 in Healthy Volunteers
Brief Title: Study of CMP-CPS-001 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CAMP4 Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPS-101
Record Dates: First submitted 2024-01-22; First posted 2024-02-08 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Antisense Oligonucleotides; Urea Cycle Disorder
MeSH Terms: conditions — Urea Cycle Disorders, Inborn

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single Ascending Dose Part (Experimental): Adult healthy volunteers in 4 cohorts of 12 will receive CMP-CPS-001 or placebo. Four dose levels will be evaluated.
  Interventions: Drug: CMP-CPS-001; Other: Placebo
- Multiple Ascending Dose Part (Experimental): Adult healthy volunteers in 4 cohorts of 12 will receive 3 monthly doses of either CMP-CPS-001 or placebo. Four dose levels will be evaluated.
  Interventions: Drug: CMP-CPS-001; Other: Placebo

INTERVENTIONS:
Drug: CMP-CPS-001 — CMP-CPS-001 consists of an antisense oligonucleotide solution that will be administered subcutaneously.
Other: Placebo — Placebo is 0.9% normal saline solution and will be administered subcutaneously.

SUMMARY:
The objective of this clinical study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple ascending doses of CMP-CPS-001 administered as a subcutaneous injection in adult healthy volunteers.

DETAILED DESCRIPTION:
This is a randomized, double-blind (Sponsor-open), and placebo-controlled study.

The SAD part will be conducted in approximately 48 healthy volunteers, in 4 cohorts of 12, randomized 3:1 to receive a single subcutaneous dose of CMP-CPS-001 or placebo. Participants will be followed for 42 days after dosing.

The MAD part will be conducted in approximately 48 healthy volunteers, in 4 cohorts of 12, randomized 3:1 to receive 3 monthly doses of CMP-CPS-001 or placebo. Participants will be followed for 56 days after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18 to 55 years inclusive at time of informed consent
* BMI ≥18.0 and ≤32 kg/m2 at screening, and ≤110 kg
* Willing and able to sign informed consent form

Exclusion Criteria:

* Any significant disease or disorder which, in the opinion of the Investigator, may either put the study participant at risk because of participation in the study, may influence the results of the study, or may affect the study participant's ability to participate in the study
* Clinically relevant illness within 7 days before the first dose of study drug
* History of intolerance to subcutaneous injection or relevant abdominal scarring
* Laboratory results outside normal ranges at screening and judged as clinically relevant by the Investigator for liver function, kidney function, and platelets
* Positive viral serology test results for human immunodeficiency virus type 1 or 2 antibodies, hepatitis B surface antigen or hepatitis C virus antibody
* Any other safety laboratory result considered clinically significant and unacceptable by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Screening (Day -36) until 42 days (SAD) or 112 days (MAD) after dosing
  Incidence of adverse events, including dose limiting toxicities, after administration of CMP-CPS-001

SECONDARY OUTCOMES:
Plasma PK | Pre-dose (Day 1) until 42 days (SAD) or 112 days (MAD) after dosing
  Plasma concentration of CMP-CPS-001
Urinary excretion of CMP-CPS-001 | 42 days (SAD) or 111 days (MAD) after dosing
  Urine concentration of CMP-CPS-001
Pharmacodynamic effect of CMP-CPS-001 on ureagenesis | Run-in (Day -8) until 42 days (SAD) or 112 days (MAD) after dosing
  Ureagenesis rate test determination

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Wong, MD, Principal Investigator — Q-Pharm Pty Ltd
Locations (1):
- Nucleus Network Brisbane (also known as Q-Pharm Pty Ltd), Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No